CLINICAL TRIAL: NCT02085122
Title: Impact of Noninvasive Ventilation With Two Levels of Pressure on Exercise Tolerance in Subjects With Heart Failure: Randomized and Controlled Clinical Trial.
Brief Title: Exercise and Noninvasive Ventilation in Heart Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Daniella Cunha Brandao, Professor Adjunto, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Larissa_ergo_vni_2
Record Dates: First submitted 2014-03-10; First posted 2014-03-12 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2013-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Noninvasive Ventilation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- noninvasive ventilation (Experimental)
  Interventions: Other: noninvasive ventilation
- Control Group (No Intervention)

INTERVENTIONS:
Other: noninvasive ventilation — Ventilatory support with bilevel positive pressure was held for 30 minutes with the volunteer sitting comfortably. A fan with two pressure levels (Vivo 40 Bi-Level, General Electric Company), which was attached to the face of the individual through a face Macara ( Respironics), was initially adopted one of 15 cmH2O IPAP and EPAP was used 5 cmH2O, making admissible pressure of 10 cm H2O, where the IPAP would be increased, subject to the comfort of the patient until the patient reached a tidal volume of 6-8 ml / kg, not exceeding the maximum of 20 cmH2O for IPAP.
  Arms: noninvasive ventilation

SUMMARY:
Introduction: Dyspnea and fatigue determine exercise intolerance in heart failure (HF) subjects, hampering performance in activities of daily living. In this context, noninvasive ventilation (NIV) has been used to minimize such impairment, increasing functional capacity Aim: To evaluate the impact of NIV on exercise performance in HF individuals. Methods: A randomized crossover clinical trial with allocation concealment consisted of two experimental phases: NIV and control, 7 days apart of each other. During NIV phase, 30 minutes of bi-level ventilation was performed. Any type of ventilator support was offered during control phase. Functional capacity was assessed by cardiopulmonary exercise test on a treadmill.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes, 18-60 years
* body mass index (BMI) <30 kg/m2
* functional class II-III according to the New York Heart Association
* of the echocardiogram últiimos 6 months showing ejection fraction (LVEF) ≤ 45% - echocardiogram of six months showing cardiac hypertrophy (left Ventricular Diastolic Diameter (LVDD)> 55mm
* Diameter Systolic left Ventricular (LVSD)> 45mm )
* optimized from the point of view of drug and (6) clinical stability

Exclusion Criteria:

* (1) unstable angina, myocardial infarction or heart surgery three months before the beginning of the research

  (2) chronic orthopedic, infectious or metabolic diseases

  (3) FEV1/FVC <70% predicted characterizing obstructive respiratory disorder; (4) active smokers

  (5) Limitation on the use of NIV: claustrophobia, inability to remain with their mouths closed, abdominal distention, hemodynamic instability, heart rate (HR) <60 bpm, recent trauma, nausea and vomiting face

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-03; Primary Completion 2013-03 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary Exercise Test | Seven days
  Cardiopulmonary exercise testing ( CPET ) was performed with symptom-limited ramp protocol (Silva et al . , 2003 ) treadmill ( Centurium 300 Micromed, Brazil ) through ErgoPC Elite ® software associated with electrocardiogram ( Micromed , Brazil ) with 12 channels . The test was performed under standard conditions of temperature, pressure and humidity ( STPD ) , breath-by - breath, being voluntary breathing in a face mask leak during exercise . Before each test the calibration of the equipment for pressure and gas volume was carried out. To ensure that patients reached the maximum effort during the examination were considered tests where patients present a respiratory exchange ratio ( R) ≥ 1.1 ( ARENA , et al 2011) .

CONTACTS AND LOCATIONS:
Locations (1):
- Departamento de Fisioterapia da UFPE, Recife, Pernambuco, Brazil

REFERENCES:
- [Result] Olson TP, Johnson BD. Influence of cardiomegaly on disordered breathing during exercise in chronic heart failure. Eur J Heart Fail. 2011 Mar;13(3):311-8. doi: 10.1093/eurjhf/hfq177. Epub 2010 Oct 16. PMID 20952768
- [Derived] Carvalho LA, Brandao DC, Campos SL, Vidal TMS, Remigio MI, Martins SM, Dornelas de Andrade A. Noninvasive Ventilation Before Maximum Exercise Test Increases Exercise Tolerance in Subjects With Heart Failure: A Crossover Study. Arch Phys Med Rehabil. 2017 May;98(5):849-855. doi: 10.1016/j.apmr.2016.09.129. Epub 2016 Oct 26. PMID 27794485
- See also: Related Info — http://www.ncbi.nlm.nih.gov/